

Version Date: 29JAN2019

Principal Investigator: Catherine J. Lee, MD

## Allogeneic Stem Cell Transplantation for Multiple Myeloma and Myelofibrosis

Lead Org. ID: HCI98381/IRB# 98381 CTO#HCI-17-HEME-07 ClinicalTrials.gov ID – NCT03303950

Principal Investigator Catherine J. Lee, MD

Blood & Marrow Transplant Program

University of Utah

2000 Circle of Hope, Rm 2152 Salt Lake City, UT 84132 Phone: (801) 587-0231

Email: Catherine.Lee@hci.utah.edu

Sub-investigator(s) Douglas Sborov, MD

Clinical Instructor, Department of Medicine

Phone: (801) 581-8394

Email: douglas.sborov@hsc.utah.edu

Vedran Radojcic, MD

Assistant Professor, Department of Medicine

Phone: (801) 213-6109

Email: vedran.radojcic@hsc.utah.edu

Daniel R. Couriel, MD, MS

Director, Blood & Marrow Transplant Program Professor,

Department of Medicine Phone: (801) 587-4056

Email: daniel.couriel@hci.utah.edu

Jo-Anna Reems, PhD (Laboratory)

Scientific Director, Cell Therapy & Regenerative Medicine Research Professor, Department of Medicine

Phone: (801) 585-6262

Email: joanna.reems@hsc.utah.edu


Principal Investigator: Catherine J. Lee, MD

Michael Boyer, MD

Associate Professor, Department of Medicine

Phone: (801) 585-3229

Email: michael.boyer@hsc.utah.edu

Josef Prchal, MD

Professor, Department of Medicine

Phone: (801) 585-3229

Email: josef.prchal@hsc.utah.edu

Tibor Kovacsovics, MD

Associate Professor, Department of Medicine

Phone: (801) 213-5621

Email: tibor.kovacsovics@hci.utah.edu

Janet Weidner, PA-C

Physician Assistant, Division of Hematology

Phone: (801) 587-0236

Email: janet.weidner@hsc.utah.edu

Mary Steinbach, DNP, APRN

Nurse Practitioner, Division of Hematology

Phone: (801) 587-1604

Email: mary.steinbach@hsc.utah.edu

Sam Shewan, PA

Physician Assistant, Division of Hematology

Phone: (801) 213-2069

Email: samuel.shewan@hsc.utah.edu

Statistician(s)

Ken Boucher

University of Utah

Huntsman Cancer Institute 2000 Circle of Hope

Salt Lake City, UT 84112

801-585-9544

kenneth.boucher@hci.utah.edu

**IND Number** 

Exempt

**Historical Protocol Versions** 

Version 1:26APR2017 Version 2:27OCT2017 Version 3: 02JUL2018

Version 4: 29JAN2019

# **TABLE OF CONTENTS**

| | <u>P</u> | age |
|---|---|---|
| LIST OI | F ABBREVIATIONS | |
| <b>PROTO</b> | COL SIGNATURE | 9 |
| <b>STUDY</b> | SUMMARY | 10 |
| OBJEC <sup>7</sup> | ΓΙVES | 12 |
| 1.1 | Primary Objectives and Endpoint | 13 |
| 1.2 | Secondary Objectives and Endpoint | |
| BACKO | GROUND | |
| 2.1 | Allogeneic in Stem Cell Transplantation in Multiple Myeloma | 13 |
| 2.2 | Allogeneic Stem Cell Transplant in Myelofibrosis | 13 |
| 2.3 | Post allograft Cyclophosphamide | 14 |
| 2.4 | Detection of minimal residual disease (MRD) following transplantation in M | ИM |
| and M | <b>1</b> F | |
| DRUG I | INFORMATION | 14 |
| 3.1 | Busulfan | 14 |
| 3.2 | Fludarabine | 15 |
| 3.3 | Cyclophosphamide | 15 |
| STUDY | DESIGN | 16 |
| 4.1 | Number of Patients | 16 |
| 4.2 | Number of Study Centers | 16 |
| 4.3 | Study Duration | |
| <b>ELIGIB</b> | ILITY CRITERIA | 17 |
| 5.1 | Inclusion Criteria | 17 |
| 5.2 | Exclusion Criteria. | 18 |
| 5.3 | Donor Inclusion Criteria | 18 |
| TREAT | MENT PLAN | 20 |
| 6.1 | Administration Schedule | |
| 6.2 | Treatment Administration | 21 |
| 6.3 | Accountability and Compliance | 22 |
| 6.4 | Prohibited Concomitant Medications | 22 |
| 6.5 | Duration of Therapy | 22 |
| TOXICI | ITIES AND DOSEAGE MODIFICATION | |
| 7.1 | Supportive Care | 23 |
| 7.2 | Diagnosis and Treatment of Acute GVHD | |
| 7.3 | Diagnosis and Treatment of Chronic GVHD | 24 |
| STUDY | CALENDAR | |
| CRITER | RIA FOR EVALUATION AND ENDPOINT | 27 |
| 9.1 | Non-relapse mortality (NRM) up to day +365 | 27 |
| 9.2 | Rate of acute GVHD grade II-IV at Day +100 post-transplant | |
| 9.3 | Cumulative chronic GVHD rates | 27 |
| 9.4 | Response (clinical and molecular, disease free survival) | |
| 9.5 | Safety | |
| 9.6 | Stopping Rules | |
| | TICAL CONSIDERATIONS | 31 |

| REGISTR. | ATION GUIDELINES | 31 |
|-----------|-----------------------------------------|----|
| DATA SU | BMISSION SCHEDULE | 31 |
| ETHICAL | AND REGULATORY CONSIDERATIONS | 32 |
| 13.1 | Informed consent | 32 |
| 13.2 | Institutional Review | 32 |
| 13.3 | Data and Safety Monitoring Plan | 32 |
| 13.4 | Adverse Events / Serious Adverse Events | 32 |
| 13.5 | SAE Reporting Requirements | 35 |
| 13.6 | Reporting of Pregnancy | |
| 13.7 | Protocol Amendments | 37 |
| 13.8 | Protocol Deviations | 37 |
| 13.9 | FDA Annual Reporting | 38 |
| 13.10 | Clinical Trials Data Bank | |
| 13.11 | Record Keeping | 38 |
| REFEREN | ICES | 38 |
| Appendice | S | 43 |

# LIST OF ABBREVIATIONS

| Abbreviation or Term <sup>1</sup> | Definition/Explanation |
|---|---|
| AE | Adverse event |
| ALT | Alanine aminotransferase |
| ANCOVA | Analysis of covariance |
| ANOVA | Analysis of variance |
| APTT | Activated partial thromboplastin time |
| AST | Aspartate aminotransferase |
| AV | Atrioventricular |
| β-HCG | Beta-human chorionic gonadotropin |
| BID | Twice daily |
| BLQ | Below limit of quantification |
| BMI | Body mass index |
| BP | Blood pressure |
| BUN | Blood urea nitrogen |
| Ca <sup>++</sup> | Calcium |
| CBC | Complete blood count |
| CFR | Code of Federal Regulations |
| CHF | Congestive heart failure |
| CI | Confidence interval |
| Cl- | Chloride |
| CLcr | Creatinine clearance |
| C <sub>max</sub> | Maximum observed concentration |
| C <sub>min</sub> | Trough observed concentration |
| CNS | Central nervous system |
| CR | Complete response |
| CRF | Case report form |
| СТ | Computed tomography |
| CTCAE | Common Toxicity Criteria for Adverse Events |

| Abbreviation or Term <sup>1</sup> | Definition/Explanation |
|---|---|
| CV | Coefficient of variation |
| CYP | Cytochrome P450 |
| D/C | Discontinue |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic case report form |
| DLT | Dose Limiting Toxicity |
| ECG | Electrocardiogram |
| Eg | Exempli gratia (for example) |
| FACS | Fluorescence Activated Cell Sorting |
| FDA | Food and Drug Administration |
| FDG-PET | Fluorodeoxyglucose (FDG)-positron emission tomography (PET) |
| GCP | Good Clinical Practice |
| GFR | Glomerular filtration rate |
| GGT | Gamma glutamyl transferase |
| GLP | Good laboratory practice |
| HBsAg | Hepatitis B surface antigen |
| HBV | Hepatitis B virus |
| HCO <sub>3</sub> - | Bicarbonate |
| HCV | Hepatitis C virus |
| HIV | Human immunodeficiency virus |
| HR | Heart rate |
| hr | Hour or hours |
| IC <sub>50</sub> | Half maximal inhibitory concentration |
| i.e. | Id est (that is) |
| IEC | Independent ethics committee |
| INR | International normalized ratio |
| IRB | Institutional review board |
| IU | International unit |

| Abbreviation or Term <sup>1</sup> | Definition/Explanation |
|---|---|
| IV | Intravenous, intravenously |
| LDH | Lactate dehydrogenase |
| LLQ | Lower limit of quantitation |
| MedRA | Medical Dictionary for Drug Regulatory Activities |
| MRI | Magnetic resonance imaging |
| MRSD | Maximum recommended starting dose |
| MTD | Maximum tolerated dose |
| NOAEL | No-observed-adverse-effect level |
| NOEL | No-observed-effect-level |
| PD | Pharmacodynamic(s) |
| PFS | Progression Free Survival |
| PK | Pharmacokinetic(s) |
| PO | Per os (administered by mouth) |
| PR | Partial response |
| PT | Prothrombin time |
| PTT | Partial thromboplastin time |
| QC | Quality control |
| RBC | Red blood cell |
| QD | Once daily |
| QTc | QT interval corrected |
| QTcF | QT interval corrected using Frederichia equation |
| SAE | Serious adverse event |
| SD | Standard deviation or stable disease |
| T <sub>1/2</sub> | Terminal elimination half-life |
| T <sub>3</sub> | Triiodothyronine |
| T <sub>4</sub> | Thyroxine |
| $T_{max}$ | Time of maximum observed concentration |
| TID | Three times daily |

| Abbreviation or Term <sup>1</sup> | Definition/Explanation |
|-----------------------------------|------------------------------------|
| TSH | Thyroid-stimulating hormone |
| ULN | Upper limit of normal |
| ULQ | Upper limit of quantitation |
| UV | Ultraviolet |
| WBC | White blood cell |
| WOCBP | Women of childbearing potential |
| WONCBP | Women of nonchildbearing potential |

All of these abbreviations may or may not be used in protocol.

Protocol name: Allogeneic Stem Cell Transplantation for Multiple Myeloma and Myelofibrosis Version Date: 29JAN2019

Principal Investigator: Catherine J. Lee, MD

## PROTOCOL SIGNATURE

I confirm that I have read this protocol, and I will conduct the study as outlined herein and according to the ethical principles stated in the latest version of the Declaration of Helsinki, the applicable ICH guidelines for good clinical practice, and the applicable laws and regulations of the federal government. I will promptly submit the protocol to the IRB for review and approval. Once the protocol has been approved by the IRB, I understand that any modifications made during the course of the study must first be approved by the IRB prior to implementation except when such modification is made to remove an immediate hazard to the subject.

I will provide copies of the protocol and all pertinent information to all individuals responsible to me who assist in the conduct of this study. I will discuss this material with them to ensure that they are fully informed regarding the study treatment, the conduct of the study, and the obligations of confidentiality.

Note: This document is signed electronically through submission and approval by the Principal Investigator at Huntsman Cancer Institute in the University of Utah IRB Electronic Research Integrity and Compliance Administration (ERICA) system. For this reason, the Principal Investigator at Huntsman Cancer Institute will not have a handwritten signature on this signature page.

# STUDY SUMMARY

| Title | A Phase II study of Allogeneic stem cell transplantation for |
|---|---|
| | multiple myeloma and myelofibrosis |
| Short Title | Allo SCT for MM and MF |
| Protocol Number | 98381 |
| IND | Exempt |
| Phase | II |
| Design | Single arm, open labeled study of allogenic stem cell |
| Design | transplantation for multiple myeloma and myelofibrosis with |
| | related and unrelated stem cell donors. |
| Study Duration | Patients will receive treatment for 2 weeks with 1 year |
| | follow up |
| | Accrual will take 3 years |
| | Total study duration will be 4 years |
| Study Center(s) | Single Center: HCI |
| Objectives | Primary endpoints: |
| | To evaluate Non-Relapse Mortality (NRM) up to day +100. |
| | Secondary endpoints: |
| | To evaluate Non-Relapse Mortality (NRM) up to day +365. |
| | To evaluate the incidence of acute GVHD and chronic GVHD up to day +365 post-transplant. |
| | To evaluate the Overall Survival and Disease Free Survival up to 1 year. |
| | To evaluate Clinical Response and Molecular Response up to 1 year. |
| Number of Subjects | 24 |
| Diagnosis and Main Eligibility | Inclusion Criteria: |
| Criteria | Age 18-75 years. |
| | ECOG status 0-1 |
| | Patients must have histologically documented Multiple Myeloma (MM) |
| | A) Patients in early relapse (less than 24 months from initiation of systemic anti-myeloma therapy which may include single or planned tandem autologous transplant) after primary therapy that included an autologous HSCT OR |


Principal Investigator: Catherine J. Lee, MD

B) Later Stage

OR

C) High risk factors defined by the presence of any one of the following detected at any time prior to enrollment: deletion of chromosome 13 by conventional cytogenetics, hypodiploidy, abnormality in chromosome 1 (1q amplification or 1p deletion), t(4;14), t(14;16), t(14;20) or deletion of 17p by fluorescence in situ hybridization (FISH) or conventional karyotyping; high risk criteria based on commercially available gene expression profiling

OR

D) extramedullary disease, plasma cell leukemia or high LDH (19)

# Patients must have histologically documented Myelofibrosis (MF)

1) Patients with DIPSS plus intermediate stage 2 or higher risk MF

OR

- 2) Subset of intermediate stage 1 patients. Defined by:
  - a) Poor-risk molecular profile (triple negative: JAK2, CALR, MPL)

OR

- b) Presence of any of the following mutations: (ASXL1, SRSF2, EZH2, IDH1/2)
  OR
- c) Severe thrombocytopenia, severe anemia, high peripheral blood blasts percentage OR
- d) Unfavorable cytogenetic abnormalities (rearrangements of chromosome 5 or 7 or  $\geq$  3 abnormalities <sup>(40)</sup>).

Principal Investigator: Catherine J. Lee, MD

| | Exclusion Criteria: |
|---|---|
| | a. Cardiac-left ventricular ejection fraction <40%, symptomatic coronary artery disease, or uncontrolled arrhythmias b. Pulmonary- FEV1 or DLCO < 40% or history of chronic use of supplemental oxygen. Temporary use of supplemental oxygen at the time of screening or registration is allowed if the investigator feels that the underlying cause of requiring oxygen is reversible by the time treatment begins c. Renal- calculated or measured GFR <30 ml/min, dialysisdependent, or history of renal transplant d. Hepatic- bilirubin > 2 X ULN, ALT> 2.5 X ULN, cirrhosis e. Patients with active or uncontrolled bacterial, viral, or fungal infections requiring systemic therapy f. Pregnant women, nursing mothers or women of childbearing potential who are unwilling to use medically accepted methods of contraception |
| Study Product, Dose, Route,<br>Regimen | Allogenic transplant using a divided regimen of busulfan at Day-5 to Day-2 and post-transplant cyclophosphamide at Day +3 and Day +4. |
| Duration of administration | 10 days |
| Reference therapy | Standard of care continuous conditioning regimen using busulfan and cyclophosphamide. |
| Statistical Methodology | Comparison of primary endpoint with historical benchmarks of patients treated with allogenic transplants. |
| | Analysis of secondary endpoints will be done descriptively. |

## **OBJECTIVES**

This study will investigate a variation on a proven conditioning program for allogeneic Hematopoietic Stem Cell Transplantation (HSCT) for treatment of patients with Multiple Myeloma (MM) and primary Myelofibrosis (PMF). The current protocol allows stem cell transplant from matched related donors (MRD), matched unrelated donors (MUD), mismatched unrelated donor(s) (mMUD) and haploidentical donor(s) (Haplo).

## 1.1 Primary Objectives and Endpoint

1.1.1 To evaluate Non-Relapse Mortality (NRM) up to day +100.

## 1.2 Secondary Objectives and Endpoint

- 1.2.1 To evaluate Non-Relapse Mortality (NRM) up to day +365.
- 1.2.2 To evaluate the incidence of acute GVHD and chronic GVHD up to day +365 post-transplant.
- 1.2.3 To evaluate the Overall Survival and Disease Free Survival up to 1 year.
- 1.2.4 To evaluate Clinical Response and Molecular Response (complete response and partial response [section 9.4]) up to 1 year

## **BACKGROUND**

The proposed conditioning regimen modifies the combination of busulfancyclophosphamide, one of the most successful in the treatment of Multiple Myeloma <sup>(2)</sup>, from a continuous conditioning regimen to a divided regimen where busulfan is given before allogeneic HSCT and cyclophosphamide on day +3 and +4 post allogeneic HSCT. This is the accepted standard therapy for Graft Versus Host Disease (GVHD) prevention in haploidentical transplantation and has been explored in the other 3 types of transplant. To allow for engraftment in this combination, a moderate dose of fludarabine is given, since busulfan alone might not be immunosuppressive enough.

This variation regimen is designed to maximize the antitumor effect in myeloma and myelofibrosis and minimizes the toxicity by PK directed busulfan administration and may also minimize acute and chronic GVHD by administering cyclophosphamide at day +3 and day +4 post allogeneic HSCT.

## 2.1 Allogeneic in Stem Cell Transplantation in Multiple Myeloma

Allogeneic HSCT is the only potentially curative therapy for Multiple Myeloma (MM). The use of reduced-intensity conditioning (RIC) has broadened the use of allogeneic HSCT in MM especially in patients with refractory disease and relapsed after an autograft. (1,2,3,4,5) B. Andersson introduced the PK directed busulfan regimen to optimize dose-targeting and reduced transplant related mortality. (6,15)

Risk criteria for allogeneic HSCT in MM are early relapse after primary therapy and/or high risk factors (i.e. cytogenetics, extramedullary disease, plasma cell leukemia or high LDH).

## 2.2 Allogeneic Stem Cell Transplant in Myelofibrosis

Allogeneic HSCT is the only curative treatment for primary myelofibrosis (PMF), a clonal myeloproliferative neoplasm with a high risk for clonal evolution and mortality.

Prognostic tools have been developed that assist in therapeutic decision making. The International Prognostic Symptom Score (IPSS) is a clinical based model to assess prognosis at the time of primary myelofibrosis diagnosis. The IPSS score was upgraded to the dynamic IPSS plus (DIPPS plus) score, which further clarified risk variables and risk categories (Appendix A) Four risk categories are included in DIPSS plus: low, intermediate 1, intermediate 2, and high. These categories are assessed by: age,

Principal Investigator: Catherine J. Lee, MD

constitutional symptoms, hemoglobin, the basis of WBC, circulating blasts, platelet count, RBC transfusions needed, and unfavorable karyotype.

Only MF patients with intermediate 2 and intermediate 1 with high risk designations according to DIPPS plus should be transplanted. (8)

## 2.3 Post allograft Cyclophosphamide

Post allograft cyclophosphamide (Cytoxan) has been introduced as measure for GVHD prevention in recipients of haploidentical, mismatched unrelated, and matched unrelated transplants. The results of post allograft cyclophosphamide are comparable to or better than other ways of immunosuppression, like ATG in mismatched and matched recipients of stem cell transplants. Post allograft cyclophosphamide is believed to work by destroying early activated donor T-cells and by sparing regulatory T-cells via increased expression of ALDH, one of the enzymes which metabolizes cyclophosphamide. (9,10,11,12,13) Post allograft cyclophosphamide as sole means of GVHD prophylaxis is not sufficient and should therefore be combined with other immunosuppressant like tacrolimus and mycophenolic acid (MMF) as standard of care.

# 2.4 Detection of minimal residual disease (MRD) following transplantation in MM and MF

Relapse represents the main cause of treatment failure after hematopoietic stem cell transplantation (HSCT). Monitoring of Minimal Residual Disease (MRD) allows for early detection and subsequent intervention prior to clinically detectable relapse.

MRD-determination will be done as a standard procedure approximately every 3-6 months in patients that achieve a complete response only.

MRD monitoring in MM is done by Flow Cytometry (preferred), ASO-PCR, by determining the VDOH rearrangements or NGS. (14,15,16)

MRD-Monitoring in MF is done by JAK2 PCR, cMPL, Calreticulin mutation PCR and donor-recipient chimerism determination.

Molecular relapse will be treated by DLI infusion (1X10<sup>6</sup>/kg BW for matched related donors as defined by the HCI BMT SOP

(https://pulse.utah.edu/policies/FilteredFor/Blood%20and%20Marrow%20Transplant. aspx – or consult with BMT pharmacist). Infusion of donor lymphocytes (DLI) leads to molecular responses in 30-50% of cases with MM and MF. (17,18)

## **DRUG INFORMATION**

## 3.1 Busulfan

For HSCT conditioning, intravenous busulfan is more often utilized due to less pharmacokinetic variability. With conditioning doses of busulfan, antiepileptic medication must be given. Seizure prophylaxis with levetiracetam should start prior to receiving busulfan and continue until at least 24 hours after the infusions are complete. Newer second-generation antiepileptics such as levetiracetam have become a favorable option due to decreased adverse effects and minimal drug interactions. Side effects of busulfan include nausea, diarrhea, myelosuppression, transient increase in liver enzymes, and rarely more serious liver and lung toxicity. (20) The pharmacokinetic levels


Principal Investigator: Catherine J. Lee, MD

of busulfan are determined by measuring levels in the blood following the first IV infusion according to HCI BMT SOPs:

#### 3.2 Fludarabine

Fludarabine or fludarabine phosphate (Fludara) is a chemotherapy drug used in the treatment of hematological malignancies (cancers of blood cells such as leukemias and lymphomas). It is a purine analog, which interferes with DNA synthesis. Fludarabine is highly effective in the treatment of chronic lymphocytic leukemia, producing higher response rates than alkylating agents, such as chlorambucil, alone. Fludarabine is used in various combinations with cyclophosphamaide, mitoxantrone, dexamethasone and rituximab in the treatment of indolent non-Hodgkins lymphomas. As part of the FLAG regiment, fludarabine is used together with cytarabine and granulocyte colony stimulating factor in the treatment of acute myeloid leukemia. Because of its immunosuppressive effects, fludarabine is also used in some conditioning regimens prior to allogeneic stem cell transplant.

## 3.3 Cyclophosphamide

Cyclophosphamide is an alkylating agent of the nitrogen mustard type (specifically, the oxazaphosphorine group). An alkylating agent adds an alkyl group to DNA. It attaches the alkyl group to the guanine base of DNA, at the number 7 nitrogen atom of the imidazole ring. This interferes with DNA replication by forming intrastrand and interstrand DNA crosslinks. Cyclophosphamide is used to treat cancers, autoimmune disorder and AL amyloidosis. As a prodrug, it is converted by liver cytochrome P450 (CYP) enzymes to form the metabolite 4-hydroxycyclophosphamide that has chemotherapeutic activity. Cyclosphosphamide has severe and life-threatening adverse effects, including acute myeloid leukemia, bladder cancer, hemorrhagic cystitis and permanent infertility, especially at higher doses. The addition of cyclophosphamide at day +3 and day +4 has two purposes: a) optimizing the antineoplastic effect against MM and MF and b) to prevent serious life-threatening GVHD.

Principal Investigator: Catherine J. Lee, MD

#### STUDY DESIGN



## Description

Patients will receive pre-transplant conditioning with busulfan (PK directed) and Fludarabine, followed by post-transplant cyclophosphamide on day +3 and day +4 as GVHD prophylaxis.

## 4.1 Number of Patients

24 patients will be enrolled. There is no limit to the ratio of MM and MF patients that enroll. (4, 8, 12 in 1<sup>st</sup>, 2<sup>nd</sup> and 3<sup>rd</sup> year)

## 4.2 Number of Study Centers

Huntsman Cancer Institute will be the sole enrolling site.

## 4.3 Study Duration

Total Study duration will be four years.

Principal Investigator: Catherine J. Lee, MD

## **ELIGIBILITY CRITERIA**

This eligibility checklist is used to determine patient eligibility and filed with investigators signature in the patient research chart.

| Patient N<br>Patient's | No<br>Init | ials: (L,F,M) |
|---|---|---|
| | | on Criteria<br>No (Response of "no" = patient ineligible) |
| 5.1.1 | | Age 18-75 years |
| 5.1.2 | | ECOG Performance status 0-1 |
| 5.1.3 | | Patients must have one of the following diagnoses of Multiple Myeloma M) or primary/secondary Myelofibrosis (MF): |
| | | Patients must have histologically documented Multiple Myeloma (MM) Appendix A. |
| | A) | Patients in early relapse (less than 24 months from initiation of systemic anti-myeloma therapy which may include single or planned tandem autologous transplant) after primary therapy that included and autologous HSCT. |
| | | OR |
| | B) | Later Stage. |
| | | OR |
| | C) | High risk factors defined by the presence of any one of the following detected at any time prior to enrollment: deletion of chromosome 13 by conventional cytogenetics, hypodiploidy, abnormality in chromosome 1 (1q amplification or 1p deletion), t(4;14), t(14;16), t(14;20) or deletion of 17p by fluorescence in situ hybridization (FISH) or conventional karyotyping; high risk criteria based on commercially available gene expression profiling. |
| | | OR |
| | D) | Extramedullary disease, plasma cell leukemia or high LDH (19). |
| | | Patients must have histologically documented Myelofibrosis (MF) Appendix A. |
| | A) | Patients with DIPSS plus intermediate stage 2 or higher risk MF. |
| | | OR |
| | B) | Subset of intermediate stage 1 patients. Defined by: |
| | | i) Poor-risk molecular profile (triple negative: JAK2, CALR, MPL). |


Principal Investigator: Catherine J. Lee, MD

#### OR

ii) Presence of any of the following mutations: ASXL1, SRSF2, EZH2, IDH1/2.

#### OR

C) Severe thrombocytopenia, severe anemia, high peripheral blood blasts percentage.

#### OR

- D) Unfavorable cytogenetic abnormalities (rearrangements of chromosome 5 or 7 or  $\geq$  3 abnormalities (40).
- 5.1.4 \_\_\_\_\_ Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

#### 5.2 Exclusion Criteria

## Yes/No (Response of "yes" = patient ineligible)

- 5.2.1 Cardiac- left ventricular ejection fraction <40%, symptomatic coronary artery disease, or uncontrolled arrhythmias.
- 5.2.2 Pulmonary- FEV1 or DLCO < 40% or history of chronic use of supplemental oxygen. Temporary use of supplemental oxygen at the time of screening or registration is allowed if the investigator feels that the underlying cause of requiring oxygen is reversible by the time treatment begins.
- 5.2.3 Renal- calculated or measured GFR <30 ml/min, dialysis-dependent, or history of renal transplant.
- 5.2.4 Hepatic- bilirubin > 2 X ULN, ALT > 2.5 X ULN or cirrhosis.
- 5.2.5 Patients with active or uncontrolled bacterial, viral, or fungal infections requiring systemic therapy.
- 5.2.6 Pregnant women, nursing mothers or women of child-bearing potential who are unwilling to use medically accepted methods of contraception
- 5.2.7 Male and female subjects not willing to agree to medically accepted methods of contraception.

## 5.3 Donor Inclusion Criteria

The evaluation of donors shall be in accordance with existing Foundation for the Accreditation of Cellular Therapy standards. The University of Utah Blood and Marrow Transplant and Myeloma Program are a FACT accredited Cellular Therapy programs.

| 5.3.1 | A related donor –fully matched. | |
|---|---|---|
| 5.3.2 | A related donor – haploidentical. | |
| 5.3.3 | An unrelated donor – fully matched. | |
| 5.3.4 | An unrelated donor $-9/10$ matched. | |
| I certify tha<br>onto this stu | at this patient meets all inclusion and exclusion criteria for enrollmenudy. | ıt |
| Investigator | r Signature Date Time | |

Principal Investigator: Catherine J. Lee, MD

#### TREATMENT PLAN

## HCI BMT SOPs found:

 $\frac{https://pulse.utah.edu/policies/FilteredFor/Blood\%20and\%20Marrow\%20Transplant.aspx}{-\ or\ consult\ with\ BMT\ pharmacist)}.$ 

## 6.1 Administration Schedule

| Therapy |
|---|
| Start Levetiracetam <sup>1</sup> (per standard of care dosing) |
| Busulfan daily dose of 3.2 mg/kg/day IV |
| Busulfan goal Css = 800 to 900 ng/mL as determined by the PI (PK Blood Draw required per HCI MBT SOPs) |
| Fludarabine 30 mg/m <sup>2</sup> IV |
| Levetiracetam |
| Busulfan |
| Fludarabine 30 mg/m <sup>2</sup> |
| Levetiracetam |
| Busulfan |
| Fludarabine 30 mg/m <sup>2</sup> |
| Levetiracetam |
| Busulfan |
| Fludarabine 30 mg/m <sup>2</sup> |
| Levetiracetam |
| Rest |
| Levetiracetam |
| HPC infusion per HCI BMT Standard of Care SOP |
| Cyclophosphamide 50mg/kg IV over 60 minutes per HCI BMT standard of Care SOP |
| Cyclophosphamide 50mg/kg IV over 60 minutes |
| Tacrolimus per standard dosing guidelines with Mycophenolate mofetil (MMF) 15 mg/kg IV or PO q8 hrs (max dose 3g/day) and continued until day +35 |

<sup>1</sup>With conditioning doses of busulfan, antiepileptic medication (levetiracetam) must be given. Seizure prophylaxis should start prior to receiving busulfan and continue at least 24 hours after the infusions are complete.

<sup>&</sup>lt;sup>2</sup>Tacrolimus and Mycophenolate mofetil (MMF) can also be used post-transplant as GVHD prophylaxis per PI discretion as HCI BMT standard of care SOP.

<sup>\*</sup>Residual or relapsing disease will be treated with DLI infusions per HCI BMT SOP.

Principal Investigator: Catherine J. Lee, MD

MF patients who take Ruxolitinib prior to transplant will continue to do so. The dose of Ruxolitinib is reduced to  $2 \times 5$  mg and continued until stable engraftment, then tapered and stopped around day +28. In case of early CMV reactivation, the drug will be tapered earlier<sup>(41)</sup>.

## 6.2 Treatment Administration

All treatments associated with protocol are commercially available agents and will be administered per institutional guidelines only to eligible patients under the supervision of the investigator or sub-investigator(s). The treatments will be prepared under the supervision of a pharmacist at Huntsman Cancer Institute. The amount of drug to be administered will be determined based on targeted PK, body surface area, ideal body weight, actual or adjusted body weight and calculated based on institutional standards.

#### 6.2.1 Busulfan:

See HCI BMT SOP for details of busulfan administration, toxicities, PK sample collection and targeted level and levetiracetam prophylaxis.

- a. Dosage: the initial dose for intravenous busulfan is 3.2 mg/kg/dose IV daily. Busulfan Css goal is 800 ng/mL to 900 ng/mL, as per the investigator's clinical judgement. Busulfan dose may need to be adjusted based on busulfan levels drawn after the first dose. Therefore, without dose adjustment, the total dose is 12.8 mg/kg. Busulfan will only be given intravenously over 3 hours from Days –5 through –2. Doses should be rounded to the nearest 1 mg.
- b. Dosage calculation is based on actual or adjusted body weight see HCI BMT SOP for calculation of chemotherapy.

#### 6.2.2 Fludarabine:

See HCI BMT SOP for details of Fludarabine administration and toxicities.

- a. Dosage: 30 mg/m²/day IV on Days -5 through Day -2, for a total dose of 120 mg/m². The dose is rounded to the nearest 5 mg and given intravenously over 30 minutes.
- b. Dosage calculation is based on actual body weight. HCI BMT SOP for calculation of chemotherapy.

Consider a 25% dose reduction of fludarabine in patients with creatinine clearance <50 mL/min. Fludarabine should be avoided in patients with creatinine clearance <30 mL/min.

#### 6.2.3 HPC infusion

Source of hematopoietic progenitor cells (HPC) to be determined by BMT attending physician. Infusion to be given per HCI BMT SOP.

## **Graft versus Host Disease prophylaxis**

## 6.2.4 Cyclophosphamide

Cyclophosphamide 50mg/kg IV over 60 minutes on Day +3 and Day +4. Post-transplant cyclophosphamide should be started between 60-72 hours after HPC


Principal Investigator: Catherine J. Lee, MD

infusion. Dosage calculation is always based on ideal body weight, unless the patient weighs less than ideal body weight, then use actual body weight.

Hydration prior to cyclophosphamide may be given according to institutional standards. Mesna should be started prior to cyclophosphamide at a dose of 100% of cyclophosphamide dose in 1 liter of 0.9% sodium chloride, given as a continuous infusion. Discontinue mesna approximately 24 hours after the last dose of cyclophosphamide.

It is crucial that no immunosuppressive agents are given until 24 hours after the completion of the post-transplant cyclophosphamide. This includes corticosteroids as anti-emetics.

#### 6.2.5 Tacrolimus

Tacrolimus will be initiated at Day +5 per standard dosing guidelines with a goal of being tapered to off by Day +180, in the absence of GVHD.

• 0.01-0.03 mg/kg/day IV continuous infusion depending on age and prophylactic antifungal choice. In some patients, tacrolimus may be started as an oral formulation at a dose of 0.045-0.06 mg/kg/dose PO BID and titrated as needed. The conversion from IV to PO tacrolimus is approximately 1:3.

## 6.2.6 Mycophenolate mofetil (MMF) WITH Tacrolimus

MMF will be initiated at Day +5 at a dose of 15mg/kg IV or PO q8 hrs (max dose 3 gm/day) and discontinued on Day +35 in the absence of GVHD.

See HCI BMT SOP for details of tacrolimus plus MMF administration:

## 6.3 Accountability and Compliance

Accountability for the treatment is the responsibility of the principal investigator. The investigator will ensure that treatment is used only in accordance with this protocol. Drug accountability records will be maintained per institutional practice.

### 6.4 Prohibited Concomitant Medications

Medications will be managed at PI discretion.

## 6.5 **Duration of Therapy**

Patients will receive a conditioning regimen, transplant, GVHD prevention and one year of assessment on study.

## TOXICITIES AND DOSEAGE MODIFICATION

This study will utilize the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0 for adverse event and serious adverse event reporting. A copy of the CTCAE Version 5.0 can be downloaded: (<a href="http://safetyprofiler-ctep.nci.nih.gov/CTC/CTC.aspx">http://safetyprofiler-ctep.nci.nih.gov/CTC/CTC.aspx</a>).

Principal Investigator: Catherine J. Lee, MD

## 7.1 Supportive Care

## 7.1.1 Prophylactic Care

All supportive measures consistent with optimal patient care will be given throughout the study. Institutional guidelines will be followed and include the following:

- Prophylactic antibiotics consisting of a quinolone or equivalent depending upon patient tolerance as per institutional standards.
- Prophylactic antifungals consisting of caspofungin, fluconazole, voriconazole, or posaconazole as per institutional standards. The use of azole antifungals should be avoided until Day +5 due to potential drug-drug interaction between azoles and cyclophosphamide.
- Prophylactic acyclovir or valacyclovir starting by day 0 and continuing until one year post transplant.
- Patients receiving haploidentical transplant, will receive filgrastim or filgrastimsndz 5 mcg/kg/day starting on Day +5 and continued until engraftment.
- Patients should be started on ursodiol prior to transplant per institutional standards. We will provide viral weekly screening for CMV and EBV as needed (see study calendar). Screening and infection treatment will be instituted per HCI BMT SOP.

## 7.2 Diagnosis and Treatment of Acute GVHD

GVHD assessment should be conducted standard of care once weekly for the first 100 days and then monthly until one year following BMT by the treating transplant physician or GVHD experienced members of the BMT team including midlevel providers using the forms provided in appendix B. Additional time points of assessment depend on clinical necessity and or when symptoms of GVHD arise.

Acute GVHD can affect various target organs, predominantly the GI tract, liver and skin. It is not defined by time of onset but by clinical symptoms. The recommended staging and grading of acute GVHD, and the functional grading of acute GVHD is presented in HCI BMT SOP (appendix B). Whenever possible, the clinical diagnosis of GVHD should be confirmed by biopsy of an affected end organ, but should not delay management. Other complications affecting the skin, liver, and gastrointestinal (GI) tract should be ruled out.

## GVHD grade I:

• topical treatment (steroid cream, tacrolimus 0.01 - 0.03%, antihistamine containing lotion against pruritus)

GVHD grade II:

- systemic treatment with corticosteroids (1mg/kg prednisolone)
   GVHD grade III and IV:
- systemic treatment with corticosteroids (2mg/kg methylprednisolone; equivalent to prednisone 2.5mg/kg) plus calcineurin inhibitor.


Principal Investigator: Catherine J. Lee, MD

For skin involvement: additional topical agents allowed. For GI tract involvement: additional nonabsorbable agents (budesonide, beclomethasone) allowed.

See HCI BMT SOP for additional treatment of acute GVHD: (<a href="https://pulse.utah.edu/policies/FilteredFor/Blood%20and%20Marrow%20Transplant.aspx">https://pulse.utah.edu/policies/FilteredFor/Blood%20and%20Marrow%20Transplant.aspx</a> – or consult with BMT pharmacist).

## 7.3 Diagnosis and Treatment of Chronic GVHD

GVHD assessments should be conducted standard of care once weekly for the first 100 days and then monthly until one year following BMT by the treating transplant physician or GVHD experienced members of the BMT team including midlevel providers.

Additional time points of assessment depend on clinical necessity and or when symptoms of GVHD arise. See HCI BMT SOP for details of chronic GVHD assessments and treatments.

Protocol name: Allogeneic Stem Cell Transplantation for Multiple Myeloma and Myelofibrosis Version Date: 29JAN2019

Principal Investigator: Catherine J. Lee, MD

# STUDY CALENDAR

| Examination | Screen ing <sup>1</sup> | Day -6 | Day<br>-5 | Day<br>-4 | Day<br>-3 | Day<br>-2 | Day<br>-1 | Day<br>0 | Day +3 | Day<br>+4 | Day<br>+28<br>M1<br>(±7<br>Days) | Day<br>+100<br>M4<br>(±7<br>Days) | Day<br>+180<br>M6<br>(±7<br>Days) | Day<br>+365<br>M12<br>(±7<br>Days) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | | | | | | , , | | | |
| Medical History | X | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | |
| Eligibility Criteria | X | | | | | | | | | | | | | |
| Disease Staging | X | | | | | | | | | | | | | |
| Pregnancy Test <sup>4</sup> | X | | | | | | | | | | | | | |
| Adverse Events <sup>7</sup> | | | | | | | | X | | | • | | | |
| Vital signs | l signs X | | X | | | | | | 2 | X | X | X | | X |
| Physical examination | X | | X | | X | 2 | X | X | X | | X | | | |
| ECOG performance status | X | | | | X | | | X | 2 | X | X | X | | X |
| CMV, EBV test | X <sup>10</sup> | | | | | | | $X^{10}$ | | | X | X | | X |
| Hematology <sup>2</sup> | X | | X | | | | | X | 2 | X | X | X | | X |
| Serum Chemistries <sup>3</sup> | X | | | | X | | | X | | X | X | X | | X |
| LDH | X | | | | | | | | | | X | X | | X |
| ЕСНО | X | | | | | | | | | | | | | X |
| Pulmonary Function Tests | X | | | | | | | | | | | | | X |
| Multiple Myeloma Disease<br>Assessments <sup>8</sup> | X | | | | | | | | | | | X | X | X |
| Myelofibrosis Disease Assessment <sup>9</sup> | X | | | | | | | | | | | X | X | X |
| Busulfan | | | X | X | X | X | | | | | | | | |
| Busulfan PK | | | X | | | | | | | | | | | |
| Fludarabine | | | X | X | X | X | | | | | | | | |
| Cyclophosphamide | | | | | | | | | X | X | | | | |


Principal Investigator: Catherine J. Lee, MD

| Transplant HSCT | | X | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Minimal Residual Disease <sup>5</sup> | X | | | | | X | X | X |
| Acute and Chronic GVHD<br>Assessment <sup>6</sup> | | | X | X | X | X | | X |
| Clinical CR up through 1 year <sup>8,9</sup> | | | | | | | X | |
| Molecular CR up through 1 year <sup>8,9</sup> | | | | | | | X | |

- 1 ALL Pre-study/Screening procedures should be completed within 4 weeks of study enrollment with the exception of laboratory tests which need to be completed within 2 weeks prior to study enrollment and bone marrow aspirate and biopsy which could be completed within 60 days of study enrollment. Prior medical history will be assessed at screening, including assessment of comorbidities.
- 2 Hematology includes CBC with differential and platelets. Assessments should be done weekly at the discretion of the investigator.
- 3 Chemistry includes Albumin, Alkaline Phosphatase, Aspartate Aminotransferase, Alanine Aminotransferase, Total Bilirubin, Calcium, Carbon Dioxide, Creatinine, Chloride, Glucose, Potassium, Protein, Sodium, Urea Nitrogen.
- 4 Pregnancy test must be done at screening for all women of childbearing potential and repeated as clinically indicated.
- 5 MRD monitoring in Multiple Myeloma done by Flow Cytometry (preferred), ASO-PCR, by determining the VDOH rearrangements or NGS. MRD-Monitoring in Myelofibrosis to be done by JAK2 PCR or cMPL or Calreticulin mutation PCR and donor-recipient chimerism determination. This testing should be done at screening to determine the molecular markers that will determine MRD after transplant. MRD-determination should be done as a standard procedure every 3-6 months ONLY if the patient has demonstrated complete response. Previous MRD testing results may be used for screening requirement, if performed within 60 days of study enrollment.
- 6 GVHD assessments for acute and chronic GVHD should be conducted as per standard of care once weekly from Day 0 to day +100. Assessments should continue monthly after day +100 until day +365.
- 7 Adverse Events will start at Day-6 and continue to Day+365.
- 8 Multiple Myeloma disease assessments should include evaluation of quantitative immunoglobulins, serum protein electrophoresis (SPEP), serum immunofixation electrophoresis (SIFE), 24-hour urine for total urine protein, urine immunofixation electrophoresis (UIFE), serum free light chains. Bone marrow aspirate and biopsy including cytogenetics, plasma cell FISH and other molecular testing for MM associated mutations and/or other chromosomal abnormalities, bone scans and/or PET/CT should be performed as clinically indicated (if supported by increased signs and symptoms). Response should be monitored every 3 6 months until disease progression.
- 9 Myelofibrosis disease assessments should include evaluation of symptoms, evaluation of the spleen by physical exam, and/or CT or MRI. Bone marrow aspirate and biopsy including cytogenetics, flow cytometry and molecular testing for MF associated mutations and/or other chromosomal abnormalities should be performed as clinically indicated (if supported by increased signs and symptoms). Response should be monitored every 3 6 months until disease progression.

10 As Needed

Principal Investigator: Catherine J. Lee, MD

#### CRITERIA FOR EVALUATION AND ENDPOINT

## 9.1 Non-relapse mortality (NRM) up to day +365

NRM is defined as death due to GVHD, infections, sepsis, organ (lung, liver, kidney) toxicity. Death from underlying disease (i.e. progression or relapse) is not considered NRM.

## 9.2 Rate of acute GVHD grade II-IV at Day +100 post-transplant

GVHD should be assessed according to the standard of care by the treating physician or other member of the BMT clinical team including mid-level providers once weekly through day +100 post transplant and monthly for 1 year. Acute GVHD may affect the skin, the gastrointestinal tract, and the liver. Diagnosis of acute GVHD is based on criteria established according to the criteria as described by the 1994 Consensus conference on acute GVHD grading. The recommended staging and grading of acute GVHD and the functional grading of acute GVHD is presented in HCI BMT SOP (see worksheet in appendix B).

#### 9.3 Cumulative chronic GVHD rates

Diagnosis of chronic GVHD is based on criteria established by the National Institutes of Health Consensus Development Project in 2005 (Filipovich et al. 2005), and recently updated in 2014. Diagnostic and distinctive manifestations of chronic GVHD are present in the skin and appendages, mouth, eyes, female genitalia, esophagus, lungs and connective tissues. Diagnosis of chronic GVHD requires the presence of at least 1 diagnostic clinical sign (e.g. poikiloderma or esophageal web) or the presence of at least 1 distinctive manifestation (e.g. keratoconjunctivitis sicca) confirmed by pertinent biopsy or other relevant tests (e.g. Schirmer test) in the same or another organs. Biopsy or other testing is not always feasible to confirm the presence of chronic GVHD and is not mandatory if the patient has at least 1 of the diagnostic findings of chronic GVHD. Other possible diagnoses for clinical symptoms must be excluded.

The National Institutes of Health Consensus Development Project recognizes 2 main categories of GVHD each of which having 2 subcategories as shown in Table 4. The broad category of chronic GVHD includes (a) classic chronic GVHD without features characteristic of acute GVHD, and (b) an overlap syndrome in which features of chronic and acute GVHD appear together.

Table 4: Categories of GVHD

| Category | Time of Symptoms after HSCT | Presence of Acute<br>GVHD Features* | Presence of Chronic GVDH Features* |
|---|---|---|---|
| Acute GVHD | | | |
| Classic acute | ≤ 100 days | Yes | No |
| Persistent, | >100 days | Yes | No |
| recurrent or late | | | |
| onset | | | |
| Chronic GVHD | | | |


Principal Investigator: Catherine J. Lee, MD

| Classic chronic | No time limit | No | Yes |
|------------------|---------------|-----|-----|
| Overlap syndrome | No time limit | Yes | Yes |

No time limit is set for the diagnosis of chronic GVHD. In the absence of histological or clinical signs or symptoms of chronic GVHD, the persistence, recurrence or new onset of characteristic skin, GI tract or liver abnormalities should be classified as acute GVHD regardless of the time of onset after transplantation.

Scoring of chronic GVHD (mild, moderate or severe) is similarly based upon criteria established by the National Institutes of Health Consensus Development Project, updated in 2014 (see worksheets appendix C). The following scoring system determines severity:

#### Mild Chronic GVHD

1 or 2 organs involved with no more than score 1

## **AND**

Lung score of 0

## **Moderate Chronic GVHD**

3 or more organs involved with no more than score 1

#### OR

At least 1 organ (not lung) with a score of 2

#### OR

Lung score 1

## **Severe Chronic GVHD**

At least 1 organ with a score of 3

## OR

Lung score of 2 or 3

## 9.4 Response (clinical and molecular, disease free survival)

A clinical and molecular response will be assessed up to Day +365.

For Multiple Myeloma, the IMWG criteria will be used to assess clinical/molecular response:

## Complete Response (CR)

Negative immunofixation on the serum and urine

#### **AND**

• Disappearance of any soft tissue plasmacytomas

## **AND**

• <5% plasma cells in bone marrow aspirates

Principal Investigator: Catherine J. Lee, MD

## **Stringent complete response (sCR)**

• Complete response as defined above plus normal FLC ratio<sup>1</sup>

#### **AND**

• Absence of clonal cells in bone marrow biopsy by immunohistochemistry ( $k/\lambda$  ration  $\leq 4:1$  or  $\geq 1:2$  for k and  $\lambda$  patients respectively after counting  $\geq 100$  plasma cells<sup>2</sup>

## **Partial Response (PR):**

- $\geq$  50% reduction of serum M-protein plus reduction in 24hr urinary M-proteins by a  $\geq$ 90% or to < 200mg per 24hr
  - o If the serum and urine M-protein are unmeasurable,
    - a ≥50% decrease in the difference between involved and uninvolved FLC levels are is required in place of the M-protein criteria
  - o If serum and urine M-proteins are unmeasurable, and serum-free light assay is also unmeasurable
    - ≥50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma-cell percentage was ≥30%.

## **AND**

If present at baseline, a  $\geq$ 50% reduction in the size (SPD)<sup>3</sup> of soft tissue plasmacytomas is also required

- 1. All recommendations regarding clinical uses relating to serum FLC levels or FLC ratio are based on results obtained with the validated Freelite test (Binding Site, Birmingham, UK).
- 2. Presence/absence of clonal cells on immunohistochemistry is based upon the  $\kappa/\lambda$  ratio. An abnormal  $\kappa/\lambda$  ratio by immunohistochemistry requires a minimum of 100 plasma cells for analysis. An abnormal ratio reflecting presence of an abnormal clone is  $\kappa/\lambda$  of >4:1 or <1:2.
- 3. Plasmacytoma measurements should be taken from the CT portion of the PET/CT, or MRI scans, or dedicated CT scans where applicable. For patients with only skin involvement, skin lesions should be measured with a ruler. Measurement of tumor size will be determined by the SPD.

## For Myelofibrosis:

## **Complete Response (CR)**

Bone marrow: Age-adjusted normocellularity; <5% blasts; ≤grade 1 MF<sup>2</sup>

## **AND**

Peripheral blood: Hemoglobin  $\ge 100$  g/L and  $\le UNL$ ; Neutrophil count  $\ge 1 \times 10^9$ /L and  $\ge UNL$ ; Platelet count  $\ge 100 \times 10^9$ /L and  $\le UNL$ ;  $\le 2\%$  immature myeloid cells<sup>3</sup>

## **AND**

Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH

## Partial Response (PR)

Peripheral blood: Hemoglobin  $\ge 100$  g/L and <UNL; Neutrophil count  $\ge 1$  x  $10^9$ /L and <UNL; Platelet count  $\ge 100$  x  $10^9$ /L and <UNL; < 2% immature myeloid cells<sup>3</sup>


Principal Investigator: Catherine J. Lee, MD

#### **AND**

Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH

## OR

Bone marrow: Age-adjusted normocellularity; < 5% blasts; ≤ grade 1 MF<sup>2</sup>

#### **AND**

peripheral blood: Hemoglobin  $\geq 85$  but  $\leq 100$  g/L and <UNL; neutrophil count  $\geq 1$  x  $10^9$ /L and <UNL; platelet count  $\geq 50$ , but  $\leq 10^9$ /L and <UNL; < 2% immature myeloid cells<sup>3</sup>

#### **AND**

Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH

EMH, extramedullary hematopoiesis (no evidence of EMH implies the absence of pathology- or imaging study-proven non-hepatosplenic EMH); LCM, left costal margin; UNL, upper normal limit.

- 1. Baseline and post-treatment bone marrow slides are to be interpreted at one sitting by a central review process. Cytogenetic and molecular responses are not required for CR assignment.
- 2. Grading of MF is according to the European classification (Thiele et al. European consensus on grading bone marrow fibrosis and assessment of cellularity. Haematologica. 2005;90:1128). It is underscored that the consensus definition of a CR bone marrow is to be used only in those patients in which all other criteria are met, including resolution of leukoerythroblastosis.
- It should also be noted that it was a particularly difficult task for the working group to reach a consensus regarding what represents a complete histologic remission.
- 3. Immature myeloid cells constitute blasts + promyelocytes + myelocytes + metamyelocytes + nucleated red blood cells. In splenectomized patients, <5% immature myeloid cells is allowed.

## 9.5 Safety

Routine safety and tolerability will be evaluated from the results of reported signs and symptoms, scheduled physical examinations, vital sign measurements, and clinical laboratory test results. More frequent safety evaluations may be performed if clinically indicated or at the discretion of the investigator.

## **Physical Examination**

Complete and symptom-directed physical examinations will be performed by a licensed physician (or physician's assistant or nurse practitioner)

## Vital Signs

Vital signs (blood pressure, respiratory rate, pulse rate and temperature) will be obtained in the sitting position.

## **Safety Laboratory Determinations**

Laboratory evaluations will be performed as noted in the flow chart.

Principal Investigator: Catherine J. Lee, MD

## 9.6 **Stopping Rules**

Stopping rules will be met when 4 out of 12 patients experience Non-relapse mortality (NRM) by Day+100. If the true probability of NRM is 50% there is an 81% chance that the trial will be stopped early for NRM. If the true probability NRM is 15% there is a 2.4% chance that the trial will be stopped early for NRM.

## STATISTICAL CONSIDERATIONS

The protocol proposes to study 24 patients with Myelofibrosis (MF) and Multiple Myeloma (MM).

The primary outcome is non relapse related mortality (NRM) for the entire cohort. The outcome will be reported along with exact binomial confidence intervals for informal comparison to the literature. A review of the literature yielded similar results for NRM in 19 studies for MM and 8 studies for MF. In MM we collected 19 studies with 1686 allogenic transplant patients and selected the 3 largest studies with 880 patients. These three studies reported NRM of 18%, 21.5%, and 22% for a weighted average of 21%. Weighted averaging revealed a benchmark of 25% for NRM. We hope to achieve a modest improvement over these results from the literature. We have 83% power to reject the null hypothesis that NRM = 25% at the one sided 0.05 significance level using an exact binomial test provided the true NRM = 6%. The null hypothesis will be rejected if  $\leq 3/24$  patients have NRM. If NRM is observed 3 or fewer out of 24 patients an exact 80% upper confidence bound will exclude 22%.

Analysis of acute and chronic GVHD and response (clinical and molecular response up to 1 year and disease free survival) is secondary and will be done descriptively. Proportions and exact binomial confidence intervals will be reported for secondary binary outcomes and Kaplan-Meier techniques will be used to report secondary time to event outcomes. Response outcomes will be reported for the entire cohort and also stratified by response to therapy prior to transplant, number of preceding treatment regimens and staging of disease at diagnosis. (21-39)

## **REGISTRATION GUIDELINES**

Patients must meet all of the eligibility requirements listed in Section 5 prior to registration.

Study related screening procedures can only begin once the patient has signed a consent form. Patients must not begin protocol treatment prior to registration.

Treatment should start within five working days after registration.

To register eligible patients on study, complete a Clinical Trials Office Patient Registration Form and submit to: <a href="mailto:CTORegistrations@hci.utah.edu">CTORegistrations@hci.utah.edu</a>.

## DATA SUBMISSION SCHEDULE

The Case Report Forms (CRFs) are a set of (electronic or paper) forms for each patient that provides a record of the data generated according to the protocol. CRF's should be created prior to the study being initiated and updated (if applicable) when amendments to the protocol are IRB approved. Data capture should be restricted to endpoints and relevant patient information required for planned manuscripts. These forms will be

Principal Investigator: Catherine J. Lee, MD

completed on an on-going basis during the study. The medical records will be source of verification of the data. During the study, the CRFs will be monitored for completeness, accuracy, legibility and attention to detail by a member of the Research Compliance Office. The CRFs will be completed by the Investigator or a member of the study team as listed on the Delegation of Duties Log. The data will be reviewed no less than annually by the Data and Safety Monitoring Committee. The Investigator will allow the Data and Safety Monitoring Committee or Research Compliance Office personnel access to the patient source documents, clinical supplies dispensing and storage area, and study documentation for the above-mentioned purpose. The Investigator further agrees to assist the site visitors in their activities.

#### ETHICAL AND REGULATORY CONSIDERATIONS

#### 13.1 Informed consent

Informed consent will be obtained from all research participants prior to performing any study procedures using the most recent IRB approved version.

## 13.2 Institutional Review

Study will be approved by the Institutional Review Board of University of Utah.

## 13.3 Data and Safety Monitoring Plan

A Data and Safety Monitoring Committee (DSMC) is established at Huntsman Cancer Institute (HCI) and approved by the NCI to assure the well-being of patients enrolled on Investigator Initiated Trials that do not have an outside monitoring review. Roles and responsibilities of the DSMC are set forth in the NCI approved plan. The activities of this committee include a quarterly review of adverse events including SAEs, important medical events, significant revisions or amendments to the protocol, and approval of cohort/dose escalations. If the DSMC and/or the PI have concerns about unexpected safety issues, the study will be stopped and will not be resumed until the issues are resolved. The DSMC also reviews and approves audit reports generated by the Research Compliance Office.

All phase II studies are reviewed by the full committee at each quarterly DSMC meeting. This includes a review of all serious adverse events (SAEs) occurring in patients treated at HCI or its affiliates as well as all grade 3 or greater toxicities for patients on treatment and within 30 day follow-up window (only if possibly, probably or definitely related).

#### 13.4 Adverse Events / Serious Adverse Events

This study will utilize the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 5.0 for AE and SAE reporting. An electronic copy of the CTCAE Version 5.0 can be downloaded from:

## http://safetyprofiler-ctep.nci.nih.gov/CTC/CTC.aspx

This is a protocol for allogeneic stem cell transplantation with the expected spectrum of transplant related SAEs like acute and chronic GVHD, life threatening infections, bleeding and graft rejection. A transplant related mortality of 10-20% is expected (2-5 patients).

Principal Investigator: Catherine J. Lee, MD

Anticipated frequent AEs during the acute transplant period (admission to day 28) are nausea, vomiting, diarrhea, fever, infections, mucositis. These will only be considered and documented as AE post engraftment

Grade 3 and 4 cytopenias will not be considered AE or SAE (as applicable) until after engraftment.

## 13.4.1 Adverse Events (AE)

An adverse event is the appearance or worsening of any undesirable sign, symptom, or medical condition occurring after starting the study drug even if the event is not considered to be related to study drug. For the purposes of this study, the terms toxicity and adverse event are used interchangeably. Medical conditions/diseases present before starting study drug are only considered adverse events if they worsen after starting study drug. Abnormal laboratory values or test results constitute adverse events only if they induce clinical signs or symptoms, are considered clinically significant, or require therapy.

Adverse event monitoring and collection will begin on Day -6 and end 365 days post-transplant. Any signs, symptoms or medical conditions occurring prior to Day -6 will be captured as medical history/baseline events. All adverse events will be captured in source documentation (with severity grading and causality noted) as defined in section 13.4; however, only events meeting the following criteria will be captured in OnCore (electronic CRFs):

- CTCAE ≥ grade 3-4 non-hematologic toxicities related to study treatment
- Relapse of the underlying hematological malignancy and acute/chronic GVHD will be documented on specific CRFs pages; this information should not be recorded on the CRF "Adverse Event" page and should not be treated as an adverse event (AE) unless leading to fatal outcome, which will trigger a SAE report (see Section 13.4.2).
- Engraftment failure needs to be documented as an AE. In case it meets SAE criteria, 13.4.2, an SAE report must be sent.

Information about all adverse events, whether volunteered by the subject, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, will be collected and recorded and followed as appropriate.

The occurrence of adverse events should be sought by non-directive questioning of the patient at each visit or phone contact during the study. Adverse events also may be detected when they are volunteered by the patient during or between visits or through physical examination, laboratory test, or other assessments. As far as possible, each adverse event should be evaluated to determine:

- 1.the severity grade based on CTCAE v.5 (grade 1-5)
- 2.its relationship to the study treatment (definite, probable, possible, unlikely, not related)
- 3.its duration (start and end dates or if continuing at final exam)
- 4.action taken (no action taken; study drug dosage adjusted/temporarily interrupted; study drug permanently discontinued due to this adverse event; concomitant


Principal Investigator: Catherine J. Lee, MD

medication taken; non-drug therapy given; hospitalization/prolonged hospitalization)

5. whether it constitutes an SAE

All adverse events will be treated appropriately. Once an adverse event is detected, it should be followed until its resolution, and assessment should be made at each visit (or more frequently, if necessary) of any changes in severity, the suspected relationship to the study treatment, the interventions required to treat it, and the outcome.

Information about common side effects already known about the study treatment is described in the Drug Information (section 3) and the FDA-approved product labels. This information will be included in the patient informed consent and will be discussed with the patient during the study as needed.

All adverse events will be immediately recorded in the patient research chart.

13.4.2 Serious Adverse Event (SAE)

Information about all serious adverse events will be collected and recorded. A serious adverse event is an undesirable sign, symptom or medical condition which:

- is fatal or life-threatening
- results in persistent or significant disability/incapacity
- is medically significant, i.e., defined as an event that jeopardizes the patient or may require medical or surgical intervention to prevent one of the outcomes listed above
- causes congenital anomaly or birth defect
- requires inpatient hospitalization or prolongation of existing hospitalization, unless hospitalization is for:
  - o routine treatment or monitoring of the studied indication, not associated with any deterioration in condition (procedures such as central line placements, paracentesis, pain control)
  - o elective or pre-planned treatment for a pre-existing condition that is unrelated to the indication under study and has not worsened since the start of study drug
  - o treatment on an emergency outpatient basis for an event not fulfilling any of the definitions of a SAE given above and not resulting in hospital admission
  - social reasons and respite care in the absence of any deterioration in the patient's general condition

The collection of SAEs will begin on Day -6 and end at Day +365.

Any death from any cause while a patient is receiving treatment on this protocol or up to 365 days post-transplant, or any death which occurs more than 365 days post-transplant but which is felt to be treatment related, must be reported.

Grade 3 and 4 cytopenias will not be considered SAE until after engraftment.

Principal Investigator: Catherine J. Lee, MD

Anticipated, but less frequent SAEs beyond day +28 are acute GVHD (liver, gut, skin), VOD, CMV activation, interstitial and fungal pneumonia, and cystitis which may require hospitalization

Anticipated, but less frequent SAEs after day +100 are, chronic GVHD, relapse of MM or MF.

If subjects fail to engraft by Day+28, this must be reported as an SAE.

Graft failure after allogenic hemaopoietic cell transplantation (AHCT) may manifest as either a lack of initial engraftment of donor cells, or loss of donor cells after minimal engraftment; this may occur for a variety of reasons, including recipient T-cells, natural killer cells, or antibodies. Risk of graft failure can be decreased by more intense conditioning, increased cell dose, or more effective immunosuppression. Occurrence of graft failure will be confirmed by the treating transplant physician.

Fatal relapses, fatal acute GVHD and fatal chronic GVHD are to be reported as SAEs.

This study should be handled like a phase II study. All phase II studies are reviewed by the full committee at each quarterly DSMC meeting. This includes a review of all serious adverse events (SAEs) occurring in patients treated at HCI as well as all grade 3 or greater toxicities for patients on treatment up to day +365 (only if possibly, probably or definitely related).

Toxicities which fall within the definitions listed above must be reported as an SAE regardless if they are felt to be treatment related or not. Toxicities unrelated to treatment that do NOT fall within the definitions above, must simply be documented as AEs in the patient research chart.

## 13.5 SAE Reporting Requirements

SAEs must be reported to the DSMC, the FDA, the IRB, according to the requirements described below:

A MedWatch 3500A form must be completed and submitted to <u>compliance@hci.utah.edu</u> within 1 business day of first knowledge or notification of event.

## **DSMC** Notifications:

- An HCI Research Compliance Officer (RCO) will process and submit the MedWatch form to the proper DSMC member as necessary for each individual study.
- The RCO will summarize and present all reported SAEs according to the Data and Safety Monitoring Plan at the quarterly DSMC meeting.

Information about all serious adverse events will be collected and recorded. A serious adverse event is an undesirable sign, symptom or medical condition which:

- is fatal or life-threatening
- results in persistent or significant disability/incapacity

Protocol name: Allogeneic Stem Cell Transplantation for Multiple Myeloma and Myelofibrosis Version Date: 29JAN2019

Principal Investigator: Catherine J. Lee, MD

- is medically significant, i.e., defined as an event that jeopardizes the patient or may require medical or surgical intervention to prevent one of the outcomes listed above
- causes congenital anomaly or birth defect
- requires inpatient hospitalization or prolongation of existing hospitalization, unless hospitalization is for:
  - o routine treatment or monitoring of the studied indication, not associated with any deterioration in condition (procedures such as central line placements, paracentesis, pain control)
  - elective or pre-planned treatment for a pre-existing condition that is unrelated to the indication under study and has not worsened since the start of study treatment
  - treatment on an emergency outpatient basis for an event not fulfilling any of the definitions of a SAE given above and not resulting in hospital admission
  - o social reasons and respite care in the absence of any deterioration in the patient's general condition

Toxicities which fall within the definitions listed above must be reported as an SAE regardless if they are felt to be treatment related or not. Toxicities unrelated to treatment that do NOT fall within the definitions above, must simply be documented as AEs in the patient research chart.

#### FDA Notifications:

- Adverse events occurring during the course of a clinical study that meet the following criteria will be promptly reported to the FDA:
- Serious
- Unexpected
- Definitely, Probably or Possibly Related to the investigational drug
- Fatal or life-threatening events that meet the criteria above will be reported within 7 calendar days after first knowledge of the event by the investigator; followed by as complete a report as possible within 8 additional calendar days.
- All other events that meet the criteria above will be reported within 15 calendar days after first knowledge of the event by the investigator.
- The RCO will review the MedWatch report for completeness, accuracy and applicability to the regulatory reporting requirements.
- The RCO will ensure the complete, accurate and timely reporting of the event to the FDA.
- The MedWatch report will be submitted to the FDA through the voluntary

Principal Investigator: Catherine J. Lee, MD

reporting method by the Regulatory Coordinator.

#### IRB Notification:

• Events meeting the University of Utah IRB reporting requirements (<a href="http://www.research.utah.edu/irb/">http://www.research.utah.edu/irb/</a>) will be submitted through the IRB's electronic reporting system within 10 working days.

#### 13.6 Reporting of Pregnancy

Although pregnancy is not considered an adverse event, it is the responsibility of investigators or their designees to report any pregnancy or lactation in a subject, including the pregnancy of a male subjects' female partner as an SAE. Pregnancies or lactation that occurs during the course of the trial or with 30 days of completing the trial or starting another new anticancer therapy, whichever is earlier, must be reported to the DSMC, IRB, FDA, and the sponsor as applicable. All subjects and female partners who become pregnant must be followed to the completion/termination of the pregnancy. Pregnancy outcomes of spontaneous abortion, missed abortion, fetal death, intrauterine death, miscarriage and stillbirth must be reported as serious events.

#### 13.7 Protocol Amendments

Any amendments or administrative changes in the research protocol during the period, for which the IRB approval has already been given, will not be initiated without submission of an amendment for IRB review and approval.

These requirements for approval will in no way prevent any immediate action from being taken by the investigator in the interests of preserving the safety of all patients included in the trial.

#### 13.8 Protocol Deviations

A protocol deviation (or violation) is any departure from the defined procedures and treatment plans as outlined in the protocol version submitted and previously approved by the IRB. Protocol deviations have the potential to place participants at risk and can also undermine the scientific integrity of the study thus jeopardizing the justification for the research. Protocol deviations are unplanned and unintentional events.

Because some protocol deviations pose no conceivable threat to participant safety or scientific integrity, reporting is left to the discretion of the PI within the context of the guidelines below. The IRB requires the **prompt reporting** of protocol deviations which are:

- Exceptions to eligibility criteria.
- Intended to eliminate apparent immediate hazard to a research participant or
- Harmful (caused harm to participants or others, or place them at increased risk of harm - including physical, psychological, economic, or social harm), or
- Possible serious or continued noncompliance

<sup>\*</sup>Medwatch 3500A form can be found online

Principal Investigator: Catherine J. Lee, MD

#### 13.9 FDA Annual Reporting

This study is IND exempt therefore there are no annual reporting requirements to the FDA.

#### 13.10 Clinical Trials Data Bank

The study will be registered on <a href="http://clinicaltrials.gov">http://clinicaltrials.gov</a> and the NCI CTRP (Clinical Trials Reporting Program) by the Clinical Trials Office.

#### 13.11 **Record Keeping**

Per 21 CFR 312.57, Investigator records shall be maintained for a period of 2 years following the date a marketing application is approved; or, if no application is filed or the application is not approved, until 2 years after the investigation is discontinued and the FDA is notified.

#### REFERENCES

- 1.) Shimoni A, Hardan I, Ayuk F, et al. Allogeneic Hematopoietic Stem-Cell Transplantation With Reduced-Intensity Conditioning in Patients With Refractory and Recurrent Multiple Myeloma. *Cancer*. 2010; 116: 3621-3630. doi: 10.1002/cncr.25228.
- 2.) Kröger N, Zabelina T, Klyuchnikov E, et al. Toxicity-reduced, myeloablative allograft followed by lenalidomide maintenance as salvage therapy for refractory/relapsed myeloma patients. *Bone Marrow Transplantation*. 2013; 48: 403-407. doi: 10.1038/bmt.2012.142.
- 3.) Patriarca F, Einsele H, Spina F, et al. Allogeneic Stem Cell Transplantation in Multiple Myeloma Relapsed after Autograft: A Multicenter Retrospective Study Based on Donor Availability. *Biol Blood Marrow Transplant*. 2012; 18: 617-626. doi: 10.1016/j.bbmt.2011.07.026.
- 4.) Holstein S, Richardson P, Laubach J, McCarthy P. Management of Relapsed Multiple Myeloma after Autologous Stem Cell Transplant. *Biol Blood Marrow Transplant*. 2015; 21: 793-798. doi: 10.1016/j.bbmt.2014.12.026.
- 5.) Kröger N, Badbaran A, Zabelina T, et al. Impact of High-Risk Cytogenetics and Achievement of Molecular Remission on Long-Term Freedom from Disease after Autologous-Allogeneic Tandem Transplantation in Patients with Multiple Myeloma. *Biol Blood and Marrow Transplant*. 2013; 19: 398-404. doi: 10.1016/j.bbmt.2012.10.008.
- 6.) Andersson BS, Madden T, Tran HT, et al. Acute Safety and pharmacokinetics of intravenous busulfan when used with oral busulfan and cyclophosphamide as pretransplantation conditioning therapy: a phase I study. *Biol Blood and Marrow Transplantation*. 2000; 6: 548-554.

doi:10.1016/S1083-8791(00)70064-4.

- 7.) Kröger N, Zabelina T, Schieder H, et al. Pilot study of reduced-intensity conditioning followed by allogeneic stem cell transplantation from related and unrelated donors in patients with myelofibrosis. *Blood.* 2009; 114: 5264-5270. doi:10.1182/blood-2009-07-234880.
- 8.) Kröger NM, Deeg JH, Olavarria E, et al. Indication and management of allogeneic stem cell transplantation in primary myelofibrosis: a consensus process by an EBMT/ELN international working group. *Leukemia*. 2015; 26(11): 2126-2133. doi: 10.1038/leu.2015.233.
- 9.) Kanakry J and Luznik L. Might haplo "be the (better) match?" *Blood*. 2016; 127: 799-800. doi:10.1182/blood-2016-01-689042.
- 10.) Gaballa S, Ge I, Fakih R, et al. Results of a 2-Arm, Phase 2 Clinical Trial Using Post-Transplantation Cyclophosphamide for the Prevention of Graft-Versus-Host Disease in Haploidentical Donor and Mismatched Unrelated Donor Hematopoietic Stem Cell Transplantation. *Cancer*. 2016: 1-11. doi: 10.1002/cncr.30180.
- Alousi A, Brammer J, Saliba R, et al. Phase II Trial of Graft-versus-Host Disease Prophylaxis with Post-Transplantation Cyclophosphamide after Reduced-Intensity Busulfan/Fludarabine Conditioning for Hematological Malignancies. *Biol Blood and Marrow Transplantation*. 2015; 21(5): 906-912. doi: 10.1016/j.bbmt.2015.01.026.
- 12.) Kröger N, Sayer H, Schwerdtfeger R, et al. Unrelated stem cell transplantation in multiple myeloma after a reduced-intensity conditioning with pretransplantation antithymocyte globulin is highly effective with low transplantation-related mortality. *Blood*. 2002; 100(2): 3919-3923. doi: 10.1182/blood-2002-04-1150.
- 13.) Moiseev I, Pirogova O, Alyanski A, et al. Graft-versus-Host Disease Prophylaxis in Unrelated Peripheral Blood Stem Cell Transplantation with Post-Transplantation Cyclophosphamide, Tacrolimus, and Mycophenolate Mofetil. *Biol Blood and Marrow Transplantation*. 2016;22(6):1037-42. doi: 10.1016/j.bbmt.2016.03.004.
- 14.) Lioznov M, Badbaran A, Fehse B, et al. Monitoring of minimal residual disease in multiple myeloma after allo-SCT: flow cytometry vs PCR-based techniques. *Bone Marrow Transplant.* 2008; 41(2008): 913-916.
- 15.) Sarasquete ME, Garcia-Sanz R, González, et al. Minimal residual disease monitoring in multiple myeloma: a comparison between allelic-specific oligonucleotide real-time quantitative polymerase chain reaction and flow cytometry. *Haematologica*. 2005; 90: 1365-1372.
- 16.) Fehse B, Chukhlovin A, Kuhlcke K, et al. Real-time quantitative Y chromosome-specific PCR (QYCS-PCR) for monitoring hematopoietic

- chimerism after sex-mismatched allogeneic stem cell transplantation. *J Hematother Stem Cell Res.* 2001; 10: 419-425.
- 17.) Klyuchnikov E, Holler E, Bornhäuser M, et al. Donor lymphocyte infusions and second transplantation as salvage treatment for relapsed myelofibrosis after reduced-intensity allografting. *Br J Haematology*. 2012; 159(2): 172-81.
- 18.) Rasche L, Röllig C, Stuher G, et al. Allogeneic Hematopoietic Cell Transplantation in Multiple Myeloma: Focus on Longitudinal Assessment of Donor Chimerism, Extramedullary Disease, and High-Risk Cytogenetic Features. *Biol of Blood and Marrow Transplant*. 2016; 22: 1988-1996.
- 19.) Giralt S, Garderet L, Durie B, et al. American Society of Blood and Marrow Transplantation, European Society of Blood and Marrow Transplantation, Blood and Marrow Transplant Clinical Trials Network, and International Myeloma Working Group Consensus Conference on Salvage Hematopoietic Cell Transplantation in Patients with Relapsed Multiple Myeloma. *Biol Blood and Marrow Transplant*. 2015; 21(12): 2039-2051. doi: 10.1016/j.bbmt.2015.09.016
- 20.) Palmer J, McCune J, Perales MA, et al. Personalizing Busulfan-Based Conditioning: Considerations from the American Society for Blood and Marrow Transplantation Practice Guidelines Committee. *Biol Blood and Marrow Transplant*. 2016; 22(11): 1915-1925. doi: 10.1016/j.bbmt.2016.07.013
- Lussana F, Rambaldi A, Finazzi MC, Et al. Allogeneic hematopoietic stem cell transplantation in patient with polycythemia vera or essential thrombocythemia transformed to myelofibrosis or acute myeloid leukemia: a report from the MPN Subcommittee of the Chronic Malignancies Working Party of the European Group for Blood and Marrow Transplantation. *Haematologica*, 2014; 99(5): 916-921. doi: 10.3324/haematol.2013.094284
- 22.) Patriarca F, Bacigalupo A, Sperotto A, et al. Allogeneic hematopoietic stem cell transplantation in myelofibrosis: the 20-year experience of the Gruppo Italiano Trapianto di Midollo Osseo (GITMO). *Haematologica*. 2008; 93(10): 1514-22. doi: 10.3324/haematol.12828
- 23.) Robin M, tabrizi R, Mohty M, et al. Allogeneic haematopoietic stem cell transplantation for myelofibrosis: a report of the Société Française de Greffe de Moelle et de Théerapie Cellulaire (SFGM-TC). *British Journal of Haematology*. 2011; 152(3): 331-339. doi: 10.111/j.1365-2141.2010.08417.x
- 24.) Rondelli D, Goldberg JD, Isola L, et al. MPD-RC 101 prospective study of reduced-intensity allogeneic hematopoietic stem cell transplantation in

Principal Investigator: Catherine J. Lee, MD

# patients with myelofibrosis. *Blood*. 2014; 124(7): 1183-91. **doi:** 10.1182/blood-2014-04-572545

- Gupta V, Malone AK, Hari PN, et al. Reduced-intensity hematopoietic cell transplantation for patients with primary myelofibrosis: a cohort analysis from the center for international blood and marrow transplant research. *Biology of Blood and Marrow Transplantation*. 2014; 20(1): 89-97. doi: 10.1016/j.bbmt.2013.10.018
- 26.) Kerbauy DMB, Gooley TA, Sale GE, et al. Hematopoietic cell transplantation as urative therapy for idiopathic myelofibrosis, advanced polycythemia vera, and essential thrombocythemia. *Biology of Blood and Marrow Transplantation*. 2007; 13(3); 355-365
- Kröger N, Holler E, Kobbe G, Bornhäuser M, et al. Allogeneic stem cell transplantation after reduced-intensity conditioning in patients with myelofibrosis: a prospective, multicenter study of the Chronic Leukemia Working Part of the European Group for Blood and Marrow Transplantation. *Blood*. 2009; 114(26):5264-70. doi: 10.1182/blood-2009-07-234880
- 28.) Ballen KK, Woolfrey AE, Zhu X, et al. Allogeneic hematopoietic cell transplantation for advanced polycythemia vera and essential thrombocythemia. *Biology Blood and Marrow Transplantation*. 2012; 18(9): 1446-1454. doi: 10.1016/j.bbmt.2012.03.009
- 29.) Gahrton G, Progress in allogeneic transplantation for multiple myeloma. *European Journal of Haematology*. 2010; 85(4): 279-289. doi: 10.1111/j.1600-0609.2010.01495.x
- 30.) Rotta M, Storer BE, Sahebi F, et al. Long-term outcome of patients with multiple myeloma after autologous hematopoietic cell transplantation and nonmyeloablative allografting. *Blood*. 2009; 113: 3383-91.
- 31.) Ayuk F, Perez-Simon JA, Shimoni A, et al. Clinical impact of human Jurkat T-cell-line-derived antithymocyte globulin in multiple myeloma patients undergoing allogeneic stem cell transplantation. *Haematologica*. 2008;93: 1343-50.
- Vesole DH, Zhang L, Flomenberg N, Greipp PR, Lazarus HM. A Phase II trial of autologous stem cell transplantation followed by mini-allogeneic stem cell transplantation for the treatment of multiple myeloma: an analysis of Eastern Cooperative Oncology Group ECOG E4A98 and E1A97. *Biol Blood Marrow Transplant*. 2009;15: 83-91.
- 33.) Crawley C, Iacobelli S, Bjorkstrand B, Apperley JF, Niederwieser D, Gahrton G. Reduced-intensity conditioning for myeloma: lower nonrelapse mortality but higher relapse rates compared with myeloablative conditioning. *Blood*. 2007; 109: 3588-94.

- 34.) Rosinol L, Perez-Simon JA, Sureda A, et al. A prospective PETHEMA study of tandem autologous transplantation versus autograft followed by reduced-intensity conditioning allogeneic transplantation in newly diagnosed multiple myeloma. *Blood.* 2008; 112-3591-3.
- 35.) Crawley C, Lalancette M, Szydlo R, et al. Outcomes for reduced-intensity allogeneic transplantation for multiple myeloma: an analysis of prognostic factors from the Chronic Leukaemia Working Party of the EBMT. *Blood*. 2005; 105:4532-9.
- Kröger N, shimoni A, Schillig G, et al. Unrelated stem cell transplantation after reduced intensity conditioning for patients with multiple myeloma relapsing after autologous transplantation. *Br J Haemtol*. 2010; 148: 323-31.
- 37.) Franssen LE, raymakers RA, Buijs A, Schmitz MF, van Dorp S, Mutis T, Lokhorst HM, van de Donk NW. Outcome of allogeneic transplantation in newly diagnosed and relapsed/refractory multiple myeloma: long-term follow-up in a single institution. *Eur J Haematol.* 2016; 97(5): 479-488. doi: 10.111/ejh.12758
- 38.) Auner HW, Szydlo R, van Biezen A, et al. Reduced intensity-conditioned allogeneic stem cell transplantation for multiple myeloma relapsing or progressing after autologous transplantation: a study by the European Group for Blood and Marrow Transplantation. *Bone marrow Transplant*. 2013; 48(11): 1395-400. doi: 10.1038/bmt.2013.73
- 39.) El-Cheikh J, Crocchiolo R, Furst S, et al. Long-term outcome after allogeneic stem-cell transplantation with reduced-intensity conditioning in patients with multiple myeloma. *Am J Hematol*. 2013; 88(5): 370-4. doi: 10.1002/ajh.23412
- 40.) Tam CS1, Abruzzo LV, Lin KI, et. al. The role of cytogenetic abnormalities as a prognostic marker in primary myelofibrosis: applicability at the time of diagnosis and later during disease course. *Blood*. 2009 Apr 30;113(18):4171-8. doi: 10.1182/blood-2008-09-178541
- 41.) Nicolaus Kröger, Sharifah Shahnaz Syed Abd Kadir et. al. Ruxolitinib during Peritransplant Period for Myelofibrosis Patients Undergoing Allogeneic Stem Cell Transplantation Reduces Acute Graft-Versus-Host Disease. Blood 2016 128:2242


Principal Investigator: Catherine J. Lee, MD

#### **APPENDICES**

#### Appendix A (staging criteria)

#### MULTIPLE MYELOMA

#### Clinical Presentation, Diagnosis and Staging

<u>High risk disease</u> — Approximately 15 percent of people with multiple myeloma have high risk disease based on cytogenetic testing (patients with translocation t (14;16)), translocation t (14;20) and deletion chromosome 17p). This is the aggressive form of multiple myeloma and may shorten survival; patients at high risk disease are treated with more aggressive therapy.

<u>Intermediate risk disease</u> — Approximately 10 percent of people with multiple myeloma have intermediate risk disease based on cytogenetic testing (patients with translocation t (4;14)). With appropriate therapy, patients with this form of multiple myeloma can have outcomes similar to those of standard risk multiple myeloma.

<u>Standard risk disease</u> — All patients with multiple myeloma who lack high or intermediate risk genetic abnormalities are considered to have standard risk multiple myeloma, and with appropriate therapy have an estimated median survival of 8 to 10 years.

#### Stage I - All of the following:

- Hemoglobin value > 10 g/dL
- Serum calcium value normal or ≤ 12 mg/dL
- Bone x-ray, normal bone structure (scale 0) or solitary bone plasmacytoma only
- Low M-component production rate (IgG value < 5 g/dL; IgA value < 3 g/dL)
- Bence Jones protein < 4 g/24 hr

#### Stage II - Neither Stage I nor Stage III

Stage III - One or more of the following:

- Hemoglobin value < 8.5 g/dL
- Serum calcium value > 12 mg/dL
- Advanced lytic bone lesions (scale 3)
- High M-component production rate (IgG value > 7 g/dL; IgA value > 5 g/dL)
- Bence Jones protein > 12 g/24 h

#### **Sub-classifications** (either A or B)

A: Relatively normal renal function (serum creatinine value < 2.0 mg/dL)

B: Abnormal renal function (serum creatinine value = 2.0 mg/dL)

The International Staging System, which is the most recent, most reliantly used risk assessment system and identifies three risk groups on the basis of serum  $\beta$ 2-microglobulin and albumin levels (Greipp et al., 2005):


Principal Investigator: Catherine J. Lee, MD

<u>Stage I</u> - Serum beta-2 microglobulin is less than 3.5 (mg/L) and the albumin level is 3.5 (g/dL) or greater

<u>Stage II</u> - Neither stage I or III, meaning that either: The beta-2 microglobulin level is between 3.5 and 5.5 (with any albumin level), OR the albumin is below 3.5 while the beta-2 microglobulin is less than 3.5

Stage III - Serum beta-2 microglobulin is 5.5 or greater.

#### **MYELOFIBROSIS**

The prognosis of MF was initially guided by the Lille score (a.k.a., the Dupriez score), which used hemoglobin and white blood cell counts to classify patients as "long-lived" (median survival of ten years) or "short-lived" (median survival of two years) (Dupriez, 1996). Patients were further grouped by risk, as shown in the table below:

| Lille risk group | Number of risk factors | Median survival (years) |
|------------------|------------------------|-------------------------|
| Low | None | 7 - 8 |
| Intermediate | 1 | 2.2 |
| High | 2 | 1 |

In the past decade the International Prognostic Scoring System (IPSS), which has been progressively updated to first the dynamic IPSS (DIPSS) and now the DIPSSplus as the understanding of the natural history and especially the impact of cytogenetics on the pathogenesis of MF has increased (Alchalby & Kroger, 2014) has gained prominence. The DIPSSplus prognostic score is based on eight risk factors (need for red blood cell transfusion, hemoglobin level, platelet count, leukocyte count, circulating blasts in the blood, constitutional symptoms, unfavorable cytogenetic profile and age). There are four risk categories based on the DIPSSplus score as show in the following table (Gangat et al., 2011):


Principal Investigator: Catherine J. Lee, MD

| Variable | IPSS | DIPSS | DIPSS plus <sup>a</sup> |
|---|---|---|---|
| Age >65 years | 1 | 1 | _ |
| Constitutional symptoms | 1 | 1 | _ |
| Hb <10 g/dL | 1 | 2 | _ |
| Leukocyte count >25×109/L | 1 | 1 | _ |
| Circulating blasts ≥1% | 1 | 1 | _ |
| Platelet count <100×109/L | - | - | 1 |
| RBC transfusion need | _ | _ | 1 |
| Unfavorable karyotype | _ | _ | 1 |
| Risk groups | IPSS risk<br>score | DIPSS<br>risk score | DIPSS plus<br>risk score <sup>b</sup> |
| Low-risk | 0 | 0 | O |
| Intermediate-1 risk | 1 | 1 or 2 | 1 |
| Intermediate-2 risk | 2 | 3 or 4 | 2 or 3 |
| High-risk | ≥3 | 5 or 6 | ≥4 |

MF – Myelofibrosis; RBC – Red blood cell; Hb – Hemoglobin; IPSS – International Prognostic Scoring System; DIPSS – Dynamic IPSS. <sup>a</sup>For DIPSS plus, the score is derived from the DIPSS score, and additional points added as per the table; <sup>b</sup>1 adverse point was assigned to DIPSS intermediate-1 risk. DIPSS intermediate-2 and high-risk were assigned 2 and 3 adverse points, respectively

Unfavorable karyotype: complex karyotype or sole or two abnormalities that include trisomy 8, 7/7q-, i(17q), 5/5q-, 12p-, inv(3), or 11q23

#### Appendix B: ACUTE GVHD GRADING SCALE

| | Acute GVHD Grading | | | |
|---|---|---|---|---|
| NAME: | | TX Date: | | |
| MRN: | | Day 100: | | |
| Week | | | Max | |
| Day | | | | |
| Date | | | | |
| | | Т | 1 | T |
| Skin | Туре | | | |
| | %BSA | | | |
| | Date | | | |
| LGI | Stool | | | |
| | Date | | | |
| UGI | Emesis | | | |
| | Date | | | |
| Liver | | | | |
| | Date | | | |
| Biops | y Date | | | |
| D' | . D lt | | | |
| вюрѕ | y Results | | | |
| GVHD | | | | |
| Treatı<br>Drug | nent, | | | |
| chang | es, | | | |
| dose<br>chang | | | | |
| start a | es,<br>and end | | | |
| dates | | | | |
| Other | | | | |
| Prepa | red By: | | Reviewed By: | |
| | | | D | |
| | | | Date/Time: | I |

| Patient Name: | | | | | Transplant Date: | |
|---|---|---|---|---|---|---|
| MRN: | | | | | Progressed to acute GVHD?: Yes / No | |
| Current GVHD Stage: | | | | | Date Progressed to aGVHD: | N/A |
| Skin: | 1 | 2 | 3 | 4 | Progressed to chronic GVHD: Yes/I | No |
| Liver: | 1 | 2 | 3 | 4 | Date Progressed to cGVHD: | N/A |
| GI: | 1 | 2 | 3 | 4 | *If primary graft failure occurs, | |
| Current Overall GVHD Grade: | | | | : | notify RCO. If acute GVHD occurs before Day +60, notify RCO: | |
| Physician Signature: | | | | | Compliance@hci.utah.edu | |
| 1 | | | | | | |



Protocol name: Allogeneic Stem Cell Transplantation for Multiple Myeloma and Myelofibrosis Version Date: 29JAN2019

Principal Investigator: Catherine J. Lee, MD

#### Clinical grading of severity of acute graft-versus-host disease

| Grade | Degree of Organ Involvement |
|---|---|
| I . | + to ++ skin rash; [and] no gut involvement; [and] no liver involvement; [and] no decrease in clinical performance |
| II | + to +++ skin rash; [or] + gut involvement [and/or] + liver involvement); [and] mild decrease in clinical performance |
| III | ++ to +++ skin rash; [and/or] ++ to +++ gut involvement [and/or] ++ to ++++ liver involvement); [and] marked decrease in clinical performance |
| IV | Similar to Grade III with ++ to ++++ organ involvement and extreme decrease in clinical performance |

# Criteria for Acute Graft-vs-Host Disease

### Clinical staging of acute graft-versus-host disease according to organ involvement.

| Stage | Skin | Liver | Intestinal Tract |
|---|---|---|---|
| 0 | No rash | Bilirubin<br>< 2.0 mg/dL<br>< 34 μmol/L | Diarrhea<br>≤500 ml/day or<br><280 ml/m²/day |
| + | Maculopapular rash <25% of body surface | Bilirubin<br>2.0 - 3.0 mg/dL<br>.34 - 52 µmol/L | Diarrhea<br>>500 but ≤1000 ml/day or<br>280-555 ml/m²/day |
| ++ | Maculopapular rash<br>25-50% of body surface | Bilirubin<br>3.1 - 6.0 mg/dL<br>53 - 103 µmol/L | Diarrhea<br>>1000 but ≤1500 ml/day or<br>556-833 ml/m²/day |
| +++ | Generalized erythroderma | Bilirubin<br>6.1 - 15.0 mg/dL<br>104 - 256 µmol/L | Diarrhea .<br>>1500 ml/day or<br>>833 ml/m²/day |
| ++++ | Generalized erythroderma<br>with bullous formation and<br>desquamation | Bilirubin<br>> 15.0 mg/dL<br>> 256 μmol/L | Severe abdominal pain with or without ileus |

### Appendix C: CHRONIC GVHD GRADING SCALE

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| PERFORMANCE SCORE: KPS ECOG LPS | Asymptomatic and<br>fully active (ECOG<br>0; KPS or LPS<br>100%) | Symptomatic,<br>fully ambulatory,<br>restricted only in<br>physically<br>strenuous activity<br>(ECOG 1, KPS<br>or LPS 80-90%) | Symptomatic,<br>ambulatory, capal<br>of self-care, >50%<br>of waking hours of<br>bed (ECOG 2,<br>KPS or LPS 60-<br>70%) | >50% of waking hours in bed (ECOG) |
| SKIN† SCORE % BSA GVHD features to be scored by BSA: Check all that apply: Maculopapular rash/erythe Lichen planus-like feature Sclerotic features Papulosquamous lesions o ichthyosis | involved<br>ema<br>s | 1-18% BSA | 19-50% BSA | >50% BSA |
| Keratosis pilaris-like GVH<br>SKIN FEATURES<br>SCORE: | No sclerotic features | | Superficial sclerotic features "not hidebound" (able to pinch) | Check all that apply: Deep sclerotic features "Hidebound" (unable to pinch) Impaired mobility Ulceration |
| Other skin GVHD features (In Check all that apply: Hyperpigmentation Hypopigmentation Poikiloderma Severe or generalized prunch Hair involvement Nail involvement Abnormality present but expenses | ritus | on-GVHD documented | cause (specify): | |
| MOUTH Lichen planus-like features present: Yes No Abnormality present but es | No symptoms | Mild symptoms with disease signs but not limiting oral intake significantly on-GVHD documented | Moderate<br>symptoms with<br>disease signs with<br>partial limitation<br>of oral intake | Severe symptoms with<br>disease signs on<br>examination with major<br>limitation of oral intake |

| olained entirely by a | Mild dry eye symptoms not affecting ADL (requirement of lubricant eye drops ≤ 3 x per day) non-GVHD documented Symptoms without significant weight | Moderate dry eye symptoms partially affecting ADL (requiring lubricant eye drops > 3 x per day or punctal plugs), WITHOUT new vision impairment due to KCS | Severe dry eye symptoms significantly affecting ADL (special eyeware to relieve pain) OR unable to work because of ocular symptoms OR loss of vision due to KCS |
|---|---|---|---|
| | Symptoms<br>without<br>significant weight | Symptoms | |
| No symptoms | without<br>significant weight | | |
| plained entirely by | loss* (<5%) non-GVHD documented | mild to moderate weight loss* (5-15%) <b>OR</b> moderate diarrhea without significant interference with daily living | with significant weight loss* >15%, requires nutritional supplement fo most calorie needs <b>OR</b> esophageal dilation <b>OR</b> severe diarrhea with significant interference with daily living |
| Normal total<br>oilirubin and<br>ALT or AP<br>< 3 x ULN | Normal total<br>bilirubin with ALT<br>≥3 to 5 x ULN or<br>AP ≥ 3 x ULN | Elevated total<br>bilirubin but<br>≤3 mg/dL or<br>ALT > 5 ULN | Elevated total<br>bilirubin > 3 mg/dL |
| plained entirely by | non-GVHD documented | cause (specify): | |
| No symptoms | Mild symptoms<br>(shortness of<br>breath after<br>climbing one flight<br>of steps) | Moderate<br>symptoms<br>(shortness of breath<br>after walking on<br>flat ground) | Severe symptoms (shortness of breath at rest; requiring $0_2$ ) |
| FEV1≥80% | FEV1 60-79% | FEV1 40-59% | FEV1 ≤39% |
| 1 | lormal total ilirubin and ALT or AP 3 x ULN blained entirely by No symptoms | lormal total Normal total ilirubin and bilirubin with ALT ≥3 to 5 x ULN or AP ≥ 3 x ULN or AP ≥ 3 x ULN blained entirely by non-GVHD documented. No symptoms Mild symptoms (shortness of breath after climbing one flight of steps) | daily living blained entirely by non-GVHD documented cause (specify): formal total Normal total Elevated total ilirubin and bilirubin with ALT bilirubin but ALT or AP $\geq 3$ to $5$ x ULN or $\leq 3$ mg/dL or $\approx 3$ x ULN AP $\geq 3$ x ULN ALT $\approx 5$ ULN blained entirely by non-GVHD documented cause (specify): No symptoms Mild symptoms (shortness of symptoms breath after (shortness of breath climbing one flight after walking on flat ground) |

Abnormality present but explained entirely by non-GVHD documented cause (specify):


Principal Investigator: Catherine J. Lee, MD

| S | CORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| P-ROM score (see below) Shoulder (1-7): Elbow (1-7): Wrist/finger (1-7): Ankle (1-4): Abnormality present but | No<br>symptoms | Mild tightness of arms or legs, normal or mild decreased range of motion (ROM) AND not affecting ADL by by non-GVHD docum | Tightness of arms or legs <b>OR</b> joint contractures, erythema thought due to fasciitis, moderate decrease ROM <b>AND</b> mild to moderate limitation of ADL ented cause (specify): | Contractures <b>WITH</b> significant decrease of ROM <i>AND</i> significant limitation of ADL (unable to tie shoes, button shirts, dress self etc.) |
| GENITAL TRACT (See Supplemental figure <sup>‡</sup> ) Not examined Currently sexually active Yes No | No signs | Mild signs <sup>‡</sup> and<br>females with or<br>without discomfort<br>on exam | Moderate signs <sup>‡</sup> and<br>may have<br>symptoms with<br>discomfort on exam | Severe signs <sup>‡</sup> with<br>or without<br>symptoms |
| Abnormality present but | explained entirel | y by non-GVHD docum | ented cause (specify): | |
| Other indicators, clinical score to severity (0-3) bas | | | | |
| Ascites (serositis) | . 7970 6 | henia Gravis | of none of man 1 | , |
| Pericardial Effusion_ | Periph | eral Neuropathy | Eosino | philia > 500/μl |
| Pleural Effusion(s) | Polym | yositis | Platelet | s <100,000/μl |
| Nephrotic syndrome_ | Weigh | nt loss>5%* without GI | symptoms Others | (specify): |
| Overall GVHD Severity<br>(Opinion of the evaluator) | □ No GV | THD Mild | ☐ Moderate | ☐ Severe |
| Photographic Range of M | Iotion (P-ROM) | | | |
| | Shoulder | 2 3 4 5<br>1 1 1 Y | 6 7(Normal) | |
| | 1 (Wors | 2 3 4 5 | 6 7 (Normal) | |
| | 1 (Worn | | 6 7(Normal) | |
| | Ankle / | 2 3 4(Normal) | | |

- † Skin scoring should use both percentage of BSA involved by disease signs <u>and</u> the cutaneous features scales. When a discrepancy exists between the percentage of total body surface (BSA) score and the skin feature score, OR if superficial sclerotic features are present (Score 2), but there is impaired mobility or ulceration (Score 3), the higher level should be used for the final skin scoring.
- \* Weight loss within 3 months.
- \*\*Lung scoring should be performed using both the symptoms and FEV1 scores whenever possible. FEV1 should be used in the final lung scoring where there is discrepancy between symptoms and FEV1 scores.

  <u>Abbreviations</u>: ECOG (Eastern Cooperative Oncology Group), KPS (Karnofsky Performance Status), LPS (Lansky Performance Status); BSA (body surface area); ADL (activities of daily living); LFTs (liver function tests); AP (alkaline phosphatase); ALT (alanine aminotransferase); ULN (normal upper limit).
- ‡ To be completed by specialist or trained medical providers (see Supplemental Figure).